CLINICAL TRIAL: NCT03475160
Title: Sildenafil Citrate for Treatment of Unexplained Recurrent Spontaneous Abortion
Brief Title: Sildenafil Citrate and Recurrent Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Walid Anwar Murad, Assistant Professor, Department of Obstetrics and Gynecology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18199
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Abortion
MeSH Terms: conditions — Abortion, Habitual | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Sildenafil Citrate (SC) vaginal suppositories compared to Placebo vaginal suppositories.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil Citrate (Active Comparator): Sildenafil Citrate vaginal suppositories: 25 mg every 6 hours. Uterine artery Doppler before treatment. Uterine artery Doppler after treatment.
  Interventions: Drug: Sildenafil Citrate vaginal suppositories; Procedure: Uterine artery Doppler before treatment; Procedure: Uterine artery Doppler after treatment
- Placebo (Placebo Comparator): Placebo vaginal suppositories: every 6 hours. Uterine artery Doppler before treatment. Uterine artery Doppler after treatment.
  Interventions: Drug: Placebo vaginal suppositories; Procedure: Uterine artery Doppler before treatment; Procedure: Uterine artery Doppler after treatment

INTERVENTIONS:
Drug: Sildenafil Citrate vaginal suppositories — Sildenafil citrate vaginal suppositories. Uterine artery Doppler before treatment. Uterine artery Doppler after treatment.
  Other Names: Sildenafil Citrate
  Arms: Sildenafil Citrate
Drug: Placebo vaginal suppositories — Placebo vaginal suppositories. Uterine artery Doppler before treatment. Uterine artery Doppler after treatment.
  Other Names: Placebo
  Arms: Placebo
Procedure: Uterine artery Doppler before treatment — Uterine artery Doppler before treatment: Uterine artery Doppler indices; PI and RI at cycle days 21-23 of the cycle preceding the pregnancy
Procedure: Uterine artery Doppler after treatment — Uterine artery Doppler after treatment: Uterine artery Doppler indices; PI and RI at the twelfth week of gestation

SUMMARY:
Two groups of unexplained recurrent spontaneous abortion, each included 65 participants. scheduled randomly into; the study group received Sildenafil Citrate and Placebo group. The intervention started from day 21-23 of the cycle preceding spontaneous pregnancy and continued till the 12th-week of gestation.

The primary outcome measure was the difference in the live birth between both groups. Secondary outcome measures were the differences between both groups regard pulsatility index (PI) and resistance index (RI), a number of take-home babies, the reported side-effects of treatment and the pregnancy-related complications.

DETAILED DESCRIPTION:
Two groups of unexplained recurrent spontaneous abortion, each included 65 participants. scheduled randomly into; the study group received Sildenafil Citrate and Placebo group. The intervention started from day 21-23 of the cycle preceding spontaneous pregnancy and continued till the 12th-week of gestation.

The primary outcome measure was the difference in the live birth between both groups. Secondary outcome measures were the differences between both groups regard PI and RI, a number of take-home babies, the reported side-effects of treatment and the pregnancy-related complications, e.g., preeclampsia and intrauterine growth restriction (|IUGR).

ELIGIBILITY:
Inclusion Criteria:

* Unexplained recurrent spontaneous abortion.

Exclusion Criteria:

* Abnormal uterine cavity.
* Luteal phase insufficiency.
* Endocrinal disorders, e.g., thyroid diseases, hyperprolactinemia, and Diabetes Mellitus.
* Antiphospholipid syndrome.
* Inherited or acquired thrombophilia.
* Patients had renal, hepatic or cardiovascular diseases, hypertension, history of smoking, treated with vasodilators or sensitive to or developed severe side-effects with Sildenafil Citrate.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
The difference between both groups in live birth | Through study completion, an average of 9 months.
  Live birth is defined as an ongoing pregnancy past to the 20th week of gestation

SECONDARY OUTCOMES:
Uterine artery PI at cycle day 21-23 preceding pregnancy | At cycle day 21-23 preceding pregnancy
  The difference between both groups regard PI at cycle day 21-23 preceding pregnancy
Uterine artery RI at cycle day 21-23 preceding pregnancy | At cycle day 21-23 preceding pregnancy
  The difference between both groups regard RI at cycle day 21-23 preceding pregnancy
Uterine artery PI at the twelfth week of gestation | At the twelfth week of gestation.
  The difference between both groups regard PI at the twelfth week of gestation
Uterine artery RI at the twelfth week of gestation | At the twelfth week of gestation.
  The difference between both groups regard RI at the twelfth week of gestation